CLINICAL TRIAL: NCT00377663
Title: Internet-Based Patient-Centered Asthma Management System
Brief Title: Internet-Based Program to Improve Asthma Management in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dimitri Christakis, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 431; R01HL079402-01A2 (NIH)
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): Participants will use the AsthmaNet web site.
  Interventions: Behavioral: AsthmaNet
- 2 (No Intervention): Participants will not use the AsthmaNet Web site.

INTERVENTIONS:
Behavioral: AsthmaNet — The AsthmaNet Web site will provide parents of children in the AsthmaNet group with individualized clinical information regarding their child's asthma care and with decision-making aids that they can share with their child's doctor. The web site will also prompt parents to make additional doctor appointments, as needed, to discuss their child's condition.
  Arms: 1

SUMMARY:
Asthma is a respiratory condition that affects millions of children. It can be controlled, however, with the proper medications and treatment. AsthmaNet, an internet-based asthma management system, aims to improve the asthma care of children by providing their parents and doctors with appropriate tools and feedback related to asthma management. The purpose of this study is to evaluate the effectiveness of AsthmaNet at improving quality of care and controlling asthma symptoms in children.

DETAILED DESCRIPTION:
In the United States, almost 9 million children have been diagnosed with asthma. It is a leading cause of hospitalization, chronic disease, and school absenteeism. With the proper treatment, most children with asthma are able to lead a normal life. However, if asthma is not adequately controlled, it can be a life-threatening disease. It is important for parents to work with their child's doctor to develop a comprehensive treatment plan that minimizes asthma symptoms. AsthmaNet, an interactive web-based system, aims to improve the quality of care for children with asthma by enhancing parents' asthma care skills and encouraging parents to discuss their child's asthma care with their doctor. AsthmaNet provides evidence-based guidelines, asthma management tools, and individually tailored feedback to both parents and physicians to improve communication and enhance asthma management skills and behaviors. The goal of this study is to evaluate the effectiveness of AsthmaNet at increasing medication and treatment adherence in children with asthma.

This 1-year study will enroll young children with asthma. Participants will be randomly assigned to either use the AsthmaNet web site or not use the web site. The web site will provide parents of children in the AsthmaNet group with individualized clinical information regarding their child's asthma care and with decision-making aids that they can share with their child's doctor. The web site will also prompt parents to make additional doctor appointments, as needed, to discuss their child's condition. All children will attend regularly scheduled doctor's appointments for asthma and receive their usual care; there are no additional study visits specifically for this study. Study researchers will review medical records to analyze medication usage and asthma symptoms. Participants in the AsthmaNet group will complete questionnaires on a monthly basis to assess asthma status; the control group will complete questionnaires at Month 6 and Year 1.

ELIGIBILITY:
Inclusion Criteria:

* Asthma
* Receives asthma care at a clinic in Western Washington
* Has access to the internet at home

Exclusion Criteria:

* Does not speak or read English

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2007-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Appropriate use of asthma controller medications | Measured at Year 1
Number of asthma symptom days | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri A. Christakis, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Christakis DA, Garrison MM, Lozano P, Meischke H, Zhou C, Zimmerman FJ. Improving parental adherence with asthma treatment guidelines: a randomized controlled trial of an interactive website. Acad Pediatr. 2012 Jul-Aug;12(4):302-11. doi: 10.1016/j.acap.2012.03.006. Epub 2012 Jun 11. PMID 22694878